CLINICAL TRIAL: NCT00225979
Title: Safety and Efficacy of Long-acting Repeatable Octreotide Acetate for Injectable Suspension vs. Surgery in Treatment-naïve Patients With Acromegaly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSMS995B2402
Record Dates: First submitted 2005-09-23; First posted 2005-09-26 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Acromegaly
Keywords: Acromegaly; Untreated; Newly diagnosed; Octreotide LAR; Pituitary surgery
MeSH Terms: conditions — Acromegaly

ARMS (1):
- SMS995 (Experimental)
  Interventions: Drug: Octreotide LAR

INTERVENTIONS:
Drug: Octreotide LAR
  Other Names: SMS995

SUMMARY:
Currently, the first line treatment for acromegaly is surgery, in order to remove the adenoma causing overproduction of growth hormone which leads to acromegaly. The objective of this study is to assess the safety and efficacy of long-acting repeatable formulation of octreotide and to compare it to the safety and efficacy of surgery in patients with acromegaly who have not had any previous treatment for acromegaly.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or previously untreated acromegalic patients
* Lack of suppression of GH nadir to <1.0 µg/L, after oral administration of 75 g of glucose (OGTT)
* IGF-I levels above the upper limits of normal, i.e. 97th percentile (adjusted for age and gender)

Exclusion Criteria:

* Requires surgery for recent significant deterioration in visual fields or other neurological signs, which are related to the pituitary tumor mass
* No evidence of pituitary adenoma on Magnetic Resonance Imaging (MRI)
* Symptomatic cholelithiasis

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2002-11; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Mean GH and IGF-I at baseline, week 12, 24 and 48

SECONDARY OUTCOMES:
Tumor volume at baseline, week 24 and 48
Signs and symptoms of acromegaly at baseline, week 12, 24 and 48
Quality of life and sleep apnea at baseline, week 12, 24 and 48
Safety and tolerability at any time on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals